CLINICAL TRIAL: NCT03179072
Title: The Impact of a Typical 8 Day Course of 'Target Weight' Driven Haemodialysis on the Hydration Status, Physical and Cognitive Function, Physical Activity and Quality of Life of Adults With End-stage Renal Disease.
Brief Title: Dehydr8 and Deactiv8
Status: Completed | Type: Observational
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government); Swansea University (Other); Bangor University (Other)
Responsible Party: Principal Investigator, Dr Zoe Saynor, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Other Study IDs: ZS001
Record Dates: First submitted 2017-05-26; First posted 2017-06-07 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Managing fluid status is a complex but fundamental part of the clinical care of people receiving haemodialysis (HD). Day-to-day fluid management is usually based on the concept of 'target weight' - the weight used to determine how much fluid should be removed during each dialysis session. However, the focus of this approach is usually on avoiding fluid overload (hypervolaemia), since this is associated with a higher incidence of cardiovascular and pulmonary events, in addition to increased morbidity and morbidity. As a consequence, a significant proportion of people on maintenance HD spend a great deal of time in a dehydrated state. Although dehydration is known to be associated with a number of unwanted consequences (e.g. headaches, severe fatigue, impaired cognitive and physiological function), there has been little research focusing on the impact dehydration has on the physical and psychosocial well-being of this patient group. Considering the short life expectancy of individuals with end-stage renal disease (ESRD) reliant on maintenance HD, particularly those who are unable to receive a renal transplant, we should be focused on improving their function and quality of life (QoL).

Key issues that need addressing prior to developing interventions in this cohort are 1) investigating the best and alternative measures to assess hydration status and 2) documenting the biopsychosocial impact of typical target weight driven HD in a well-designed study.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) represents the final common pathway for all progressive renal disease. As of December 2014, 58,968 people in the UK were receiving renal replacement therapy (RRT), of which almost half were receiving maintenance haemodialysis (HD; UK Renal Registry Report (2014)). The Wessex Kidney Centre cares for ~1,600 patients receiving RRT, of which >700 receive HD. The median age of our cohort is 66.7 years, similar to that of all incident UK-based patients in 2014 (64.5 years). The RRT recipient population is however growing and, increasingly, patients are more elderly with comorbidities. These individuals are unlikely to receive transplantation and will therefore depend on dialysis indefinitely. Optimising their quality of life (QoL) should be a priority.

Currently, a standard HD prescription includes a specific volume of ultrafiltration, set to achieve a clinically derived estimate of 'target weight'. Acutely, hypervolaemia (fluid overload) can be life threatening, whilst chronically it is associated with hypertension and an increased cardiovascular risk. Accordingly, target weight is typically prescribed to allow for interdialytic weight gains. The sequential reduction of target weight to achieve the lowest possible target weight (dry weight probing), thought to improve blood pressure (BP) control, left ventricular mass index and long-term outcomes, is favoured by many nephrologists. However, this results in dehydration and is associated with increased intradialytic symptoms, including intradialytic hypotension, which itself brings an increased risk of cardiac death. Local data from the Wessex Kidney Centre suggests that patients experiencing a greater drop in systolic BP pre- to post-dialysis are more likely to experience symptomatic hypotension during dialysis. Intradialytic BP variability is also detrimental to long-term outcomes. Achieving ideal hydration is therefore important for not only reducing symptomatology, but also improving BP control and cardiovascular health in these patients. Poor cardiovascular health contributes to the reduced physical function characterising this group, which along with physical (in)activity is associated with a poorer prognosis in this patient group. Furthermore, increased rates of depression and cardiovascular disease have been associated with poor physical function in this group.

There is, however, little research documenting how dehydration impacts individuals undergoing dialysis. Specifically, few studies have assessed the link between (de)hydration and frailty, although better physical function has been associated with a higher pre-dialysis BP, which may simply reflect better hydration. Experience from the Wessex Kidney Centre suggests that dehydrated dialysis patients suffer from increasing intradialytic symptomatology and a prolonged dialysis recovery time, during which they complain of prolonged fatigue. However, no studies have documented whether improving the hydration of dialysis patients improves not only their intra- and interdialytic symptomatology, but also their physiological/cognitive function, fatigue, physical (in)activity and, ultimately, QoL. Establishing the relationships between dehydration and these outcomes is essential, since hydration status can be easily and rapidly adjusted. One reason there is limited research in this area is that hydration status of individuals undergoing dialysis is difficult to objectively assess, which itself warrants further investigation.

ELIGIBILITY:
Inclusion Criteria:

The participant must meet ALL of the following criteria to be considered eligible for the study:

* Male or female > 18 years of age with ESRD and on maintenance HD for > 3 months
* Haemoglobin > 10 mg/dL
* Participant is willing and able to give informed consent for participation in the study
* Participant can understand and cooperate with the study protocol

Exclusion Criteria:

The participant may not enter the study if ANY of the following criteria apply:

* Haemoglobin ≤ 10 mg/dL
* Unable to understand or cooperate with the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with end-stage renal disease receiving in-hospital haemodialysis at the Wessex Kidney Centre will be invited to participate. This centre cares for ~700 HD patients, of which ~120 receive in-hospital HD three times a week. As more males have ESRD, it is likely that we will have a higher proportion of males. Participant's clinical records will remain at the hospital as usual.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
HHYDRATION STATUS - Change in saliva osmolality following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in saliva osmolality (BIA), sit-to-stand changes in heart rate, thirst perception scale
Hydration status - Change in plasma osmolality following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in plasma osmolality
Hydration status - Change in bioelectrical impedance analysis following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in bioelectrical impedance analysis
Hydration status - change in saliva flow rate following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in saliva flow rate
Thirst perception - Change in thirst perception following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in simple rating on visual analogue scale
Physical function - change in physical function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in muscular endurance (heel rises)
Physical function - change in physical function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in muscular endurance (30-seconds sit-to-stand)
Physical function - change in physical function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in muscular endurance (toe lifts)
Physical function - change in physical function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in fine motor skills (Moberg's picking-up test)
Physical function - Change in physical function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in muscle strength (handgrip strength)
Physical function - change in physical function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in endurance and walking capacity in patients capable of doing so (6 minute walk test).
Cognitive function - change in cognitive function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis (day 8)
  Change from baseline in cognitive function - KDQoL Questionnaire
Cognitive function - change in cognitive function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), pre-dialysis (day 3), pre-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change from baseline in cognitive function - EQ-5D-5L Questionnaire
Cognitive function - change in cognitive function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Post-dialysis (day 1), similar time of day (day 2), post-dialysis (day 3), similar time of day (day 4), post-dialysis (day 5), similar time of day (day 6), similar time of day (day 7), post-dialysis (day 8)
  Change from baseline in cognitive function - EQ-5D-5L Questionnaire (part 2 repeated only)
Physical Activity following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Continuous for 8 day period
  Accelerometry (hip mounted)
Physical Activity - change in physical activity across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), pre-dialysis (day 8)
  Change from baseline in physical activity - Rapid Assessment of Physical Activity (RAPA) Questionnaire
Sleep quality following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Continuous during 8 days (sleep diary each morning)
  Accelerometry / sleep diary

SECONDARY OUTCOMES:
Assessment of acceptability | Following involvement with the study (within 1 week)
  Semi-structured interviews will be used to examine the acceptability of alternative markers of hydration status. Specifically, interviews will explore research methods, and physical and cognitive function, PA, and QoL. Approximately 15-20 semi-structured interviews will be necessary to reach a point of data saturation where no new information is provided.
Haemodynamic function - change in haemodynamic function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change in blood pressure
Haemodynamic function - change in haemodynamic function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Change in ScvO2 - measured in those who dialyse through a central venous catheter
Haemodynamic function - change in haemodynamic function following a single session of haemodialysis (short-term) and across typical 8 days of treatment (longer-term) | Baseline (day 1: pre-dialysis 1), post-dialysis 1 (day 1), pre-dialysis (day 3), post-dialysis (day 3), pre-dialysis (day 5), post-dialysis (day 5), pre-dialysis (day 8), post-dialysis (day 8)
  Changes in resting heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD, until all avenues of further funding have been exhausted.